CLINICAL TRIAL: NCT02285673
Title: Efficacy of Umbilical Cord Mesenchymal Stem Cells in Duchenne Muscular Dystrophy: Phase 1/2 Study
Brief Title: Efficacy of Umbilical Cord Mesenchymal Stem Cells in Duchenne Muscular Dystrophy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Ercument Ovali, Specialist, Haematology, Acibadem University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DMD-UC-MSC-1
Record Dates: First submitted 2014-11-05; First posted 2014-11-07 (Estimated); Last update posted 2014-11-07 (Estimated); Status verified 2014-11

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: umbilical cord, mesenchymal stem cell
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Umbilical Cord Mesenchymal Stem Cell (Experimental)
  Interventions: Biological: Umbilical Cord Mesenchymal Stem Cell

INTERVENTIONS:
Biological: Umbilical Cord Mesenchymal Stem Cell
  Other Names: umbilical cord mesenchymal stem cells

SUMMARY:
Duchenne muscular dystrophy (DMD) is a genetic disorder caused by an absence of dystrophin and characterized by progressive muscle degeneration. There is no cure for DMD at present but, there are several strategies under-researched for treatment of DMD such as steroid treatment, gene theraphy, exon skipping, stop codon read through and gene repair, cell theraphy and theraphy with drug that help to produce utrophin protein.

The aim of this study is investigate the eficacy of human umblical cord mesenchymal stem cells on DMD and understanding if wild type gene can be transfered to the patient.

ELIGIBILITY:
Inclusion Criteria:

- Patients with diagnosis of DMD that is proven clinically and genetically Age between 7-20 Patients need partial respiratory support, during the day Patients have less than or equal to stage I NIH, Liver, renal and cardiac function Patients without cancer Patients without allergic disease Patients without bleeding diathesis,

Exclusion Criteria:

Patients need complete respiratory support Patients have more than to stage II NIH, Liver, renal and cardiac function Patients have bleeding diathesis and allergic disease

Ages: 7 Years to 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-02 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Duchenne muscular dystrophy gene expression | up to 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- Acibadem Labcell, Istanbul, Uskudar, Turkey (Türkiye)

REFERENCES:
- [Background] Lapidos KA, Kakkar R, McNally EM. The dystrophin glycoprotein complex: signaling strength and integrity for the sarcolemma. Circ Res. 2004 Apr 30;94(8):1023-31. doi: 10.1161/01.RES.0000126574.61061.25. PMID 15117830
- [Background] Miller JB, Schaefer L, Dominov JA. Seeking muscle stem cells. Curr Top Dev Biol. 1999;43:191-219. doi: 10.1016/s0070-2153(08)60382-8. PMID 9891887
- [Background] Cirak S, Arechavala-Gomeza V, Guglieri M, Feng L, Torelli S, Anthony K, Abbs S, Garralda ME, Bourke J, Wells DJ, Dickson G, Wood MJ, Wilton SD, Straub V, Kole R, Shrewsbury SB, Sewry C, Morgan JE, Bushby K, Muntoni F. Exon skipping and dystrophin restoration in patients with Duchenne muscular dystrophy after systemic phosphorodiamidate morpholino oligomer treatment: an open-label, phase 2, dose-escalation study. Lancet. 2011 Aug 13;378(9791):595-605. doi: 10.1016/S0140-6736(11)60756-3. Epub 2011 Jul 23. PMID 21784508
- [Background] Mendell JR, Rodino-Klapac LR, Sahenk Z, Roush K, Bird L, Lowes LP, Alfano L, Gomez AM, Lewis S, Kota J, Malik V, Shontz K, Walker CM, Flanigan KM, Corridore M, Kean JR, Allen HD, Shilling C, Melia KR, Sazani P, Saoud JB, Kaye EM; Eteplirsen Study Group. Eteplirsen for the treatment of Duchenne muscular dystrophy. Ann Neurol. 2013 Nov;74(5):637-47. doi: 10.1002/ana.23982. Epub 2013 Sep 10. PMID 23907995
- [Background] Goemans NM, Tulinius M, van den Akker JT, Burm BE, Ekhart PF, Heuvelmans N, Holling T, Janson AA, Platenburg GJ, Sipkens JA, Sitsen JM, Aartsma-Rus A, van Ommen GJ, Buyse G, Darin N, Verschuuren JJ, Campion GV, de Kimpe SJ, van Deutekom JC. Systemic administration of PRO051 in Duchenne's muscular dystrophy. N Engl J Med. 2011 Apr 21;364(16):1513-22. doi: 10.1056/NEJMoa1011367. Epub 2011 Mar 23. PMID 21428760
- [Background] Kerkis I, Ambrosio CE, Kerkis A, Martins DS, Zucconi E, Fonseca SA, Cabral RM, Maranduba CM, Gaiad TP, Morini AC, Vieira NM, Brolio MP, Sant'Anna OA, Miglino MA, Zatz M. Early transplantation of human immature dental pulp stem cells from baby teeth to golden retriever muscular dystrophy (GRMD) dogs: Local or systemic? J Transl Med. 2008 Jul 3;6:35. doi: 10.1186/1479-5876-6-35. PMID 18598348